CLINICAL TRIAL: NCT03181360
Title: Tenecteplase in Wake-up Ischaemic Stroke Trial (TWIST). A Randomised-controlled Trial of Thrombolytic Treatment With Tenecteplase for Acute Ischaemic Stroke Upon Awakening
Brief Title: Tenecteplase in Wake-up Ischaemic Stroke Trial
Acronym: TWIST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of North Norway (Other)
Collaborators: UiT The Arctic University of Norway (Other); The Royal Norwegian Ministry of Health (Other); Norwegian Health Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/1070/REC North; 2014-000096-80 (EudraCT Number)
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Ischemic Stroke; Stroke, Acute
Keywords: ischemic stroke; wake-up; thrombolysis; tenecteplase; computed tomography
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tenecteplase (Active Comparator): Tenecteplase + Best standard treatment
  Interventions: Drug: Tenecteplase
- Control (Other): No tenecteplase + Best standard treatment
  Interventions: Other: Control

INTERVENTIONS:
Drug: Tenecteplase — Single dose intravenous injection of recombinant fibrin-specific tissue plasminogen activator (tenecteplase) 0.25 mg (200 IU) per kg body weight up to a maximum of 25 mg (5000 IU), given as a bolus over approx. 10 seconds.
  Other Names: Metalyse
  Arms: Tenecteplase
Other: Control — Best standard treatment
  Arms: Control

SUMMARY:
Stroke is a leading causes of death and disability. At least 20% of strokes occur during sleep, so- called 'wake up stroke'. Thrombolysis with the clot-busting drug alteplase is effective for acute ischaemic stroke, provided that it is given within 4.5 hours of symptom onset. Patients with wake-up stroke are currently ineligible for clot-busting therapy. Previous studies indicate that many wake-up strokes occur just before awakening.

In this study, patients with wake-up stroke will be randomized to thrombolysis with tenecteplase and best standard treatment or to best standard treatment without thrombolysis. Tenecteplase has several potential advantages over alteplase, including very rapid action and that it can be given as a single injection. Prior to thrombolysis, a brain scan must be done to exclude bleeding or significant brain damage as a result from the stroke. We will use a CT scan to inform this decision. CT is used as a routine examination in all stroke patients. Other studies testing clot-busting treatment in wake-up stroke are using alteplase and more complex brain scans, which are not routinely available in the emergency situation in all hospitals.

DETAILED DESCRIPTION:
Background:

One in five strokes occur during sleep, but patients with "wake-up" stroke are not given thrombolytic therapy because time of stroke onset is unknown. On-going trials are testing alteplase, and use MRI techniques for selection of patients. Tenecteplase has many pharmacological advantages over alteplase: greater fibrin specificity, very rapid action, longer half-life, and single bolus administration. In addition, patient selection based on MRI findings risks excluding many patients that might otherwise benefit. TWIST will test tenecteplase and will not use MRI techniques for selection of patients. Plain CT and CT angiography (if possible) will be performed before randomisation, and CT perfusion will be performed at selected centres, as part of a sub-study.

Study design: TWIST is an international, multi-centre, randomised, open-label, blinded-endpoint trial of tenecteplase for acute ischaemic 'wake-up' stroke.

Study questions:

1. Can tenecteplase given <4.5 hours of awakening improve functional outcome at 3 months?
2. Can findings on cerebral plain CT and CT angiography (and CT perfusion, at selected centres) identify patients who benefit from such treatment, compared to other patients?

Patients eligible for treatment who are able to receive tenecteplase within 4.5 hours of waking, will be randomly allocated to treatment with tenecteplase in addition to best standard treatment, versus best standard treatment.

Randomisation and treatment: Central randomisation (over the internet) to tenecteplase 0.25 mg/mg i.v. (maximum dose 25 mg) plus best medical treatment vs. best medical treatment alone.

Imaging: All patients will undergo CT and CT angiography (CTA, if possible) before randomisation and on day 2. CT perfusion (CTP) will be performed at selected centres, as part of a sub-study.

Follow-up and primary effect variable: Centralised follow-up via telephone or mail at 3 months. The primary effect variable is functional outcome (modified Rankin Scale score).

Study size and centers: 600 patients from centers in Norway, Sweden, Denmark, Finland, Estonia, Latvia, Lithuania, United Kingdom, Switzerland and New Zealand.

ELIGIBILITY:
Inclusion Criteria:

* Stroke symptoms on awakening that were not present before sleep
* Clinical diagnosis of stroke with limb weakness with NIHSS score >=3, or dysphasia
* Treatment with tenecteplase is possible within 4.5 hours of awakening
* Written consent from the patient, non-written consent from the patient (witnessed by non-participating health care personnel), or written consent from the nearest family member

Exclusion Criteria:

* Age <18 years
* NIHSS score >25 or NIHSS consciousness score >2, or seizures during stroke onset
* Findings on plain CT that indicate that the patient is unlikely to benefit from treatment:

  * Infarction comprising more than >1/3 of the middle cerebral artery territory on plain CT or CT perfusion
  * Intracranial haemorrhage, structural brain lesions which can mimic stroke (e.g cerebral tumour)
* Active internal bleeding of high risk of bleeding, e.g.:

  * Major surgery, trauma or gastrointestinal or urinary tract haemorrhage within the previous 21 days, or arterial puncture at a non-compressible site within the previous 7 days
  * Any known defect in coagulation, e.g. current use of vitamin K antagonist with an INR >1.7 or prothrombin time >15 seconds, or use of direct thrombin inhibitors or direct factor Xa inhibitors during the last 24 hours (unless reversal of effect can be achieved by agents such as idarucizumab) or with elevated sensitive laboratory tests (such as activated partial thromboplastin time (aPTT), international normalized ratio (INR), platelet count, ecarin clotting time, thrombin time (TT), or appropriate factor Xa activity assays), or heparins during the last 24 hours or with an elevated aPTT greater than the upper limit of normal
  * Known defect of clotting or platelet function or platelet count below 100,000/mm3 (but patients on antiplatelet agents can be included)
  * Ischaemic stroke or myocardial infarction in previous 3 months, previous intracranial haemorrhage, severe traumatic brain injury or intracranial or intraspinal operation in previous 3 months, or known intracranial neoplasm, arteriovenous malformation or aneurysm
* Contraindications to tenecteplase, e.g., acute bacterial endocarditis or pericarditis; acute pancreatitis; severe hepatic dysfunction, including hepatic failure, cirrhosis, portal hypertension; active hepatitis; systemic cancer with increased bleeding risk; haemostatic defect including secondary to severe hepatic, renal disease; organ biopsy; prolonged cardiopulmonary resuscitation > 2 min (within 2 weeks)
* Persistent blood pressure elevation (systolic ≥185 mmHg or diastolic ≥110 mmHg), despite blood pressure lowering treatment
* Blood glucose <2.7 or >20.0 mmol/L (use of finger-stick measurement devices is acceptable)
* Pregnancy, positive pregnancy test, childbirth during last 10 days, or breastfeeding. In any woman of childbearing potential, a pregnancy test must be performed and the result assessed before trial entry
* Other serious or life-threatening disease before the stroke: severe mental or physical disability (e.g. Mini Mental Status score <20, or mRS score ≥3), or life expectancy less than 12 months
* Patient unavailability for follow-up (e.g. no fixed address)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional outcome at 3 months. | 3 months
  Functional outcome will be assessed by the modified Rankin Scale (mRS), values 0-6

SECONDARY OUTCOMES:
Symptomatic intracranial haemorrhage during the first 7 days. | First 7 days
  1. Symptoms (neurological deterioration, new headache, new acute hypertension, new nausea or vomiting, or sudden decrease in conscious level).
  2. Intracranial haemorrhage on brain MRI or CT.
Asymptomatic intracranial haemorrhage during the first 7 days. | First 7 days
  Intracranial haemorrhage on brain MRI or CT without: neurological deterioration, new headache, new acute hypertension, new nausea or vomiting or sudden decrease in consciousness level.
Recurrent ischaemic stroke during the first 7 days | First 7 days
  Neurological deterioration (increase of ≥2 on NIHSS, after exclusion of other causes for neurological deterioration) occurring after 72 hours will be considered as a recurrent stroke. A recurrent stroke will be classified as ischaemic if imaging has excluded haemorrhage.
Death from all cause | First 7 days
  Death will be classified according to cause:
  1. Initial stroke
  2. Recurrent stroke
  3. Myocardial infarction
  4. Pneumonia
  5. Other
Death from all cause | 3 months
  Death will be classified according to cause:
  1. Initial stroke
  2. Recurrent stroke
  3. Myocardial infarction
  4. Pneumonia
  5. Other
Barthel Index score | 3 months
  Ordinal scale for measuring performance in activities of daily living
EuroQol Score (EQ-5D) | 3 months
  Measure of health-related quality of life
Mini Mental State Examination | 3 months
  30-point questionnaire for measurement of cognitive impairment
Health-economic variables | 3 months
  Costs related to length of hospital stay, nursing home care after discharge, re-hospitalisations during first 3 months
Functional outcome at 3 months | 3 months
  Functional outcome assessed by dichotomized mRS; values 0-1 vs 2-6.

CONTACTS AND LOCATIONS:
Overall Officials: Ellisiv B Mathiesen, Principal Investigator — University Hospital of North Norway
Locations (83):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States
- Denmark (2):
  - Bispebjerg hospital, Copenhagen
  - Odense University Hospital, Odense
- Estonia (4):
  - Pärnu Hospital, Pärnu
  - East Tallin Central Hospital, Tallinn
  - West Tallin Central Hospital, Tallinn
  - Tartu University Clinic, Tartu
- Finland (5):
  - Satakunta Central Hospital, Pori, Satakunta
  - Helsinki University Hospital, Helsinki
  - Siun sote - Joint municipal authority for North Karelia social and health services, Joensuu
  - Pohjois-Kymen sairaala, Kouvola
  - Central Hospital in Vaasa, Vaasa
- Riga East University Hospital, Riga, Latvia
- Lithuania (5):
  - Alytus S. Kudirkos Hospital, Alytus
  - Lithuanian University of Health Sciences Kauno Klinikos, Kaunas
  - Klaipeda Seamen's Hospital, Klaipėda
  - Republican Vilnius University Hospital, Vilnius
  - Vilnius University Hospital, Vilnius
- Christchurch Hospital, Christchurch, New Zealand
- Norway (19):
  - Sørlandet sykehus HF Arendal, Arendal
  - Ålesund sjukehus Helse Møre og Romsdal, Ålesund
  - Drammen sykehus Vestre Viken HF, Drammen
  - Sørlandet Sykehus HF Flekkefjord, Flekkefjord
  - Helse Førde HF, Førde
  - Nordlandssykehuset Lofoten Gravdal, Gravdal
  - Helse Finnmark Hammerfest, Hammerfest
  - University Hospital of North Norway, Harstad, Harstad
  - Helse Finnmark HF Kirkenes, Kirkenes
  - Sørlandet sykehus Kristiansand HF, Kristiansand
  - Sykehuset Levanger, Levanger
  - Akershus universitetssykehus (Ahus), Lørenskog
  - Helgelandssykehuset Mosjøen, Mosjøen
  - University Hospital of North Norway, Narvik, Narvik
  - Bærum sykehus Vestre Viken HF, Sandvika
  - Sykehuset Telemark Skien, Skien
  - Stavanger Universitetssjukehus, Stavanger
  - University Hospital of North Norway, Tromsø, Tromsø
  - St Olavs Hospital, Trondheim
- Sweden (11):
  - Ängelholm Hospital, Ängelholm
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Hässleholm Sjukhus, Hässleholm
  - Central Hospital Karlstad, Karlstad
  - Skåne University Hospital Lund, Lund
  - Skåne University Hospital Malmö, Malmo
  - Skaraborg Hospital Skövde, Skövde
  - Karolinska sjukhuset, Solna
  - Saint Göran Hospital, Stockholm
  - Danderyd Hospital, Stockholm
  - Akademiska Sjukhuset, Uppsala
- Switzerland (2):
  - University Hospital Basel, Basel
  - Groupement Hospitalier Ouest Lémanique, Nyon
- United Kingdom (32):
  - Pinderfields Hospital, Wakefield, Mid Yorkshire
  - Northumbria Specialist Emergency Care Hospital, Cramlington, Northumberland
  - Aberdeen Royal Infirmary, Aberdeen
  - Arrowe Park, Birkenhead
  - University Hospital Birmingham, Birmingham
  - Royal Bournemoth and Christchurch Hospital, Bournemouth
  - Addenbrookes Hospital, Cambridge
  - Countess of Chester Hospital NHS Foundation Trust, Chester
  - University Hospitals Coventry & Warwickshire, Coventry
  - Royal Derby Hospital, Derby
  - Royal Infirmary of Edinburgh Hospital, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Gloucestershire Royal Hospital, Gloucester
  - Calderdale Royal Infirmary, Halifax
  - Hull University Teaching Hospital, Hull
  - Leeds General Infirmary, Leeds
  - Leicester Royal Infirmary, Leicester
  - Royal Liverpool University Hospital, Liverpool
  - University College London, London
  - King´s College Hospital, London
  - St Georges Hospital, London
  - Charing Cross Hospital, London
  - Royal London Hospital, London
  - Luton and Dunstable University Hospital, Luton
  - Morriston Hospital, Morriston
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - Salford Royal Hospital, Salford
  - Southhampton General Hospital, Southampton
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Musgrove Park Hospital, Taunton
  - Yeovil District Hospital, Yeovil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roaldsen MB, Eltoft A, Wilsgaard T, Christensen H, Engelter ST, Indredavik B, Jatuzis D, Karelis G, Korv J, Lundstrom E, Petersson J, Putaala J, Soyland MH, Tveiten A, Bivard A, Johnsen SH, Mazya MV, Werring DJ, Wu TY, De Marchis GM, Robinson TG, Mathiesen EB; TWIST Investigators. Safety and efficacy of tenecteplase in patients with wake-up stroke assessed by non-contrast CT (TWIST): a multicentre, open-label, randomised controlled trial. Lancet Neurol. 2023 Feb;22(2):117-126. doi: 10.1016/S1474-4422(22)00484-7. Epub 2022 Dec 19. PMID 36549308
- [Derived] Eltoft A, Wilsgaard T, Roaldsen MB, Soyland MH, Lundstrom E, Petersson J, Indredavik B, Putaala J, Christensen H, Korv J, Jatuzis D, Engelter ST, De Marchis GM, Werring DJ, Robinson T, Tveiten A, Mathiesen EB. Statistical analysis plan for the randomized controlled trial Tenecteplase in Wake-up Ischaemic Stroke Trial (TWIST). Trials. 2022 May 19;23(1):421. doi: 10.1186/s13063-022-06301-0. PMID 35590386
- [Derived] Roaldsen MB, Lindekleiv H, Eltoft A, Jusufovic M, Soyland MH, Petersson J, Indredavik B, Tveiten A, Putaala J, Christensen H, Korv J, Jatuzis D, Engelter ST, Marco De Marchis G, Wilsgaard T, Werring DJ, Robinson T, Mathiesen EB, Berge E. Tenecteplase in wake-up ischemic stroke trial: Protocol for a randomized-controlled trial. Int J Stroke. 2021 Oct;16(8):990-994. doi: 10.1177/1747493020984073. Epub 2021 Jan 14. PMID 33446083

DOCUMENTS (1):
  • Study Protocol (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/60/NCT03181360/Prot_001.pdf